CLINICAL TRIAL: NCT00912015
Title: A Comparison of the Analgesic Efficacy and Safety of Once Daily Tramadol OAD Tablets to Twice Daily Tramadol BID for the Treatment of Osteoarthritis of the Knee (Extension Protocol) and Open Label Safety Follow-Up
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Labopharm Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDT3-001-E1-A1; NCT00912015 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2009-04-09; First posted 2009-06-03 (Estimated); Results first posted 2009-06-03 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Pain; Osteoarthritis, Knee
MeSH Terms: conditions — Pain; Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Tramadol OAD 200mg (Experimental)
  Interventions: Drug: Tramadol OAD
- Tramadol OAD 300mg (Experimental)
  Interventions: Drug: Tramadol OAD
- Tramadol OAD 400mg (Experimental)
  Interventions: Drug: Tramadol OAD
- Tramadol OAD 100mg (Other): Despite provision in the protocol that the minimum daily dose was 200 mg, 2 patients took 100 mg against instructions.
  Interventions: Drug: Tramadol OAD 100mg

INTERVENTIONS:
Drug: Tramadol OAD
  Arms: Tramadol OAD 200mg
Drug: Tramadol OAD
  Arms: Tramadol OAD 300mg
Drug: Tramadol OAD
  Arms: Tramadol OAD 400mg
Drug: Tramadol OAD 100mg
  Arms: Tramadol OAD 100mg

SUMMARY:
The purpose of this study is to evaluate the long-term safety (up to one year) of Tramadol Once-A-Day (OAD) tablets at the highest doses: 200-400 mg

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female patients between the ages of 40-75 with a diagnosis of Osteoarthritis of the knee consistent with the ACR Clinical Classification Criteria for Arthritis of the Knee (Altman, R. et al., 1991):

   * Current knee pain,
   * Less than 30 minutes of morning stiffness with or without crepitus on active motion.
   * Confirmation either by arthroscopy or radiologist's report (X-rays showing osteophytes, joint space narrowing or subchondral bone sclerosis {eburnation}) within one year prior to entry into the study.
2. ESR < 40 mm/hour
3. WOMAC Pain Subscales total score of more than or equal to 150 mm at baseline.
4. Oral and written language comprehension at a level sufficient to comply with the protocol and complete study-related materials.
5. The Patient has signed and dated the REB approved, written, informed consent prior to study participation.

Exclusion Criteria:

1. Known rheumatoid arthritis or any other rheumatoid disease.
2. Secondary arthritis, i.e. any of the following: septic arthritis; inflammatory joint disease; gout; pseudogout; Paget's disease; joint fracture; acromegaly; fibromyalgia; Wilson's disease; Ochronosis; Haemochromatosis; Osteochondromatosis; heritable arthritic disorders; or collagen gene mutations.
3. Obesity Class II (BMI more than or equal to 35) (NIH, 2000)
4. Major illness requiring hospitalization during the 3 months before commencement of the screening period.
5. Unwillingness to cease taking medication other than the study medication for arthritic pain, any other concomitant pain, or OA medications.
6. Patients who have previously failed tramadol HCl therapy or those who discontinued tramadol HCl due to adverse events.
7. Patients who are taking or within the last 3 weeks have taken the following medications: monoamine oxidase inhibitors; tricyclic antidepressants and other tricyclic compounds (e.g. cyclobenzaprine, promethazine); neuroleptics; selective serotonin reuptake inhibitors; or other drugs which reduce seizure threshold.
8. Patients who are taking or have taken another investigational agent within the last 30 days.
9. Patients with a history of seizure disorder other than Infantile Febrile Seizures.
10. Patients who are opioid dependent.
11. Patients with bowel disease causing malabsorption.
12. Patients who are pregnant or lactating or patients of child-bearing potential who are unwilling to utilize a medically approved method of contraception during participation in this clinical trial.
13. Patients with significant liver disease, defined as active hepatitis or elevated liver enzymes >3 times the upper boundary of the normal range.
14. Patients with significant renal disease, defined as creatinine clearance <30 mL/min as estimated by the method of Levey et al., 1999.
15. Current substance abuse or dependence, other than nicotine.
16. Allergy or adverse reaction to tramadol or any structurally similar drugs e.g. opiates.
17. Any other condition that, in the opinion of the investigators, would adversely affect the patient's ability to complete the study or its measures.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2002-03; Primary Completion 2003-07 (Actual); Study Completion 2003-07 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Tramadol OAD 200mg: All Patients who Received 1x200 mg Tramadol OAD Tablet daily for at Least 350 days.
  OAD = Once-A-Day.
- Tramadol OAD 300mg: All Patients who Received 1x300 mg Tramadol OAD Tablet daily for at Least 350 days.
  OAD = Once-A-Day.
- Tramadol OAD 400mg: All Patients who Received 1x400 mg Tramadol OAD Tablet daily for at Least 350 days.
  OAD = Once-A-Day.
- Tramadol OAD 100mg: All Patients who Received 1x100 mg Tramadol OAD Tablet daily for at Least 350 days.
  OAD = Once-A-Day.
Period: Overall Study
Arm/Group | Tramadol OAD 200mg | Tramadol OAD 300mg | Tramadol OAD 400mg | Tramadol OAD 100mg
Started | 141 (Dose at which a patient spent the longest time.) | 70 (Dose at which a patient spent the longest time.) | 25 (Dose at which a patient spent the longest time.) | 2 (Two patients took 100 mg against instructions in protocol that the minimum daily dose was 200 mg.)
Completed | 125 | 62 | 22 | 0
Not Completed | 16 | 8 | 3 | 2
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 8 | 3 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 1
Not completed — Adverse Event | 6 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tramadol OAD 200mg | Tramadol OAD 300mg | Tramadol OAD 400mg | Tramadol OAD 100mg | Total
Number analyzed (Participants) | 141 | 70 | 25 | 2 | 238
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 87 | 42 | 16 | 2 | 147
  >=65 years | 54 | 28 | 9 | 0 | 91
Age Continuous [Mean (Standard Deviation); unit: years] | 60.1 (9.3) | 60.5 (8.8) | 58.5 (10.8) | 56.0 (5.7) | 60.0 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 58 | 21 | 1 | 203
  Male | 18 | 12 | 4 | 1 | 35

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events: 12-months Safety Population
Description: Spontaneous adverse events were recorded for patients who received the same dose for at least 350 days. A treatment emergent adverse event (TEAE) was associated to the dose level on which a patient was 2 days prior to the TEAE. Only TEAEs which could be associated with the dose level on which the patient was for the longest time were considered.
Time Frame: 12 months
Population: Patients who received the same dose for at least 350 days (12 months)
Measure: Number; unit: participants
Arm/Group | Tramadol OAD 200mg | Tramadol OAD 300mg | Tramadol OAD 400mg | Tramadol OAD 100mg
Number analyzed (Participants) | 43 | 24 | 8 | 0
participants
  Constipation | 14 | 9 | 1 |
  Dizziness | 9 | 0 | 0 |
  Nausea | 10 | 4 | 1 |
  Somnolence | 6 | 2 | 0 |
  Headache | 7 | 5 | 2 |

ADVERSE EVENTS:
Arm/Group | Tramadol OAD 200mg | Tramadol OAD 300mg | Tramadol OAD 400mg | Tramadol OAD 100mg
Serious Adverse Events (participants affected / at risk) | 4/141 | 1/70 | 1/25 | 0/2
Other Adverse Events (participants affected / at risk) | 74/141 | 34/70 | 8/25 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tramadol OAD 200mg (N=141) | Tramadol OAD 300mg (N=70) | Tramadol OAD 400mg (N=25) | Tramadol OAD 100mg (N=2)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carcinoid Tumour NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular Disorder NOS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Essential Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tramadol OAD 200mg (N=141) | Tramadol OAD 300mg (N=70) | Tramadol OAD 400mg (N=25) | Tramadol OAD 100mg (N=2)
Abdominal pain upper (Gastrointestinal disorders) | 5 (6) | 4 (4) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 26 (62) | 16 (33) | 2 (3) | 1 (8)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 26 (45) | 8 (11) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 11 (14) | 4 (4) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 4 (5) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 14 (20) | 8 (13) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 34 (61) | 10 (20) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (6) | 1 (2) | 0 (0) | 1 (2)
Somnolence (Nervous system disorders) | 26 (51) | 8 (15) | 1 (1) | 1 (2)
Sweating increased (Skin and subcutaneous tissue disorders) | 5 (6) | 2 (2) | 2 (2) | 0 (0)
Weakness (General disorders) | 10 (16) | 6 (8) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submitting results communications, the investigator shall allow Labopharm at least 30 days to review the proposed communication. If the proposed publication/disclosure risks Labopharm's ability to patent any invention related to the study, the publication or disclosure will be modified or delayed to allow Labopharm to seek patent protection. This statement does not give Labopharm any editorial rights other than to restrict the disclosure of Labopharm's confidential information.